CLINICAL TRIAL: NCT04559828
Title: Attenuation of Inflammatory Processes Associated With Alzheimer's Disease After Consumption of Pomace Olive Oil.
Acronym: ORIVA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Javier Sánchez Perona, Tenured Scientist, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 20191185 ORIVA
Record Dates: First submitted 2020-09-09; First posted 2020-09-23 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pomace olive oil (Active Comparator): 50 g of pomace olive oil will be administered in a single dose together with a breakfast composed of 3 slices of whole-grain bread, 5 g of tomato pureé and 200 ml of milk.
  Interventions: Other: Experimental meal
- High-oleic sunflower oil (Active Comparator): 50 g of high-sunflower oil will be administered in a single dose together with a breakfast composed of 3 slices of whole-grain bread, 5 g of tomato pureé and 200 ml of milk.
  Interventions: Other: Experimental meal

INTERVENTIONS:
Other: Experimental meal — Two dietary oils will be administrated as part of a single experimental meal, for the present is a postprandial phase study.

SUMMARY:
Alzheimer's disease (AD) is the most common cause of dementia and its prevalence will multiply in the coming years, so it is urgent to establish preventive and therapeutic measures. AD it is characterized by cerebrovascular and parenchymal accumulation of protein deposits enriched in amyloid-beta (Aβ) as a consequence of alterations of the blood-brain barrier. More than 60% of plasma Aβ is associated with triglyceride-rich lipoproteins (TRL), being higher in subjects with AD. Microglia act as resident macrophages and play a crucial role in most neuropathologies, since it is activated after homeostasis impairment in the brain, and surrounds amyloid plaques in patients with AD. As a result of microglial activation, a large number of pro-inflammatory markers are released, mediated by alterations in the redox state, through the generation of ROS by the complex NADPH oxidase.

In a previous study, the investigators demonstrated in BV-2 cells that artificial TRL are capable of activating microglia and trigger an inflammatory process. In addition, the investigators showed that some of lipophilic minor components of pomace olive oil simultaneously modulate oxidative stress and the inflammatory response in microglia. The investigators suggested that these results should be replicated in humans after consumption of pomace olive oil.

Therefore, in the present study we formulate the hypothesis that human TRL are capable of activating microglia and that such activation can be attenuated when those particles are generated after consumption of pomace olive oil. The results of the study would lay the foundation for the start of clinical trials demonstrating the effect of pomace oil in reducing the risk of development and progression of AD.

DETAILED DESCRIPTION:
In a previous study, the investigators demonstrated that triglyceride-rich lipoproteins (TRL), which transport dietary lipid components, are able of activating microglia, which could be associated with the state of neuroinflammation in patients of Alzheimer's disease. In addition, the investigators also demonstrated that some of the minor fat-soluble components of olive pomace oil simultaneously modulate oxidative stress and the inflammatory response in microglia, so that these components could have the ability to protect the brain from microglial overactivation when transported in TRL.

In that study, the investigators used artificial TRL that were manufactured ad-hoc in the laboratory, in order to be able to test the effect of the compounds both individually and together. Now is the time to consolidate the results using human TRL, obtained after the consumption of olive pomace oil. The investigators expect that the results of this study will reveal that the intake of olive pomace oil can prevent the release of inflammatory markers caused by the overactivation of microglia, which could be associated to a reduction in the risk of development and progression of Alzheimer's disease.

Objectives and design

To test this hypothesis, two specific objectives will be addressed:

1. To obtain and characterize human TRL obtained after the intake of olive pomace oil.
2. To evaluate the mitigating effect of the microglial activation by TRL obtained after the intake of olive pomace oil.

The study has been designed as a randomized and crossover trial in the postprandial phase in healthy subjects, which will be divided into two groups to which a pomace oil and high-oleic sunflower oil will be administered.

Activities

The specific objectives set out in the project will be addressed through the execution of the activities that are detailed below:

1. Selection of volunteers and administration of olive pomace oil. 1.1. Obtaining and characterizing the experimental oils. 1.2. Recruitment and selection of volunteers. 1.3. Clinical trial in the postprandial phase.
2. Isolation and characterization of human TRL. 2.1. General determinations in blood serum. 2.2. Characterization of TRL.
3. Microglial activation in cells treated with human TRL. 3.1. Assays in cell cultures. 3.2. Analytical determinations. 3.3. Data processing and reporting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals.
* Subjects will be recruited after a complete biochemical and haematological analysis yields results within normal limits

Exclusion Criteria:

* Digestive or metabolic conditions.
* Overweight or obesity.
* Intolerance to food components or ingredients.
* Any condition affecting lipid metabolism.
* Any inflammatory condition.
* Habitual drug intake of any kind.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Inflammation markers | Postprandial (6 hours)
  Release of proinflammatory markers TNF-α, IL-6 and IL-1β by BV2 cells treated with TRL obtained after the intake of pomace olive oil or high-oleic sunflower oil.

SECONDARY OUTCOMES:
Redox markers | Postprandial (6 hours)
  Concentrations of the redox markers reactivo oxygen species and total and reduced glutathione in BV2 cells treated with TRL obtained after the intake of pomace olive oil or high-oleic sunflower oil.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de la Grasa (IG-CSIC), Seville, Spain

IPD SHARING:
Plan to Share IPD: No